CLINICAL TRIAL: NCT02360280
Title: Intravenous Sub-anesthetic Ketamine Treatment in Treatment-Resistant Depression
Brief Title: Efficacy of Repeated Ketamine Infusions for Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Mayo Clinic (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNA-018-14S
Record Dates: First submitted 2015-01-29; First posted 2015-02-10 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Treatment-resistant Depression
Keywords: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Six ketamine infusions (Experimental): Six infusions of 0.5 mg/Kg of ketamine hydrochloride solution over 2 weeks.
  Interventions: Drug: ketamine
- Single ketamine infusion preceded by 5 midazolam infusions (Active Comparator): Single infusion of 0.5 mg/Kg of ketamine hydrochloride solution preceded by midazolam 0.045 mg/kg over 2 weeks.
  Interventions: Drug: ketamine; Drug: midazolam

INTERVENTIONS:
Drug: ketamine — sedative
Drug: midazolam — sedative
  Arms: Single ketamine infusion preceded by 5 midazolam infusions

SUMMARY:
About one-third of depressed patients will not get better after multiple antidepressant treatments. This situation put a high burden on patients with depression due to worsening quality of life and increasing health care costs. Difficult-to-treat depression might be even worse among Veterans given that the frequency of depressive symptoms is 2 to 5 times higher than among the general US population. A breakthrough discovery happened in recent years when investigators found that one infusion from an old anesthetic named ketamine showed high efficacy and rapid antidepressant effect (sometimes within hours) but lasted only up to a week. The investigators propose to study if multiple infusions of ketamine can provide greater and longer antidepressant effects than one infusion. If that is the case, multiple infusions could be an alternative to relieve depressive symptoms that do not response to multiple antidepressant drugs.

DETAILED DESCRIPTION:
Recent studies have found rapid and highly efficacious antidepressant effects of a single ketamine infusion in treatment-resistant depression (TRD). However, a single infusion appears insufficient to maintain response as most patients return to previous depressive state within a week. The strategy of multiple infusions to increase efficacy and sustain antidepressant effects has not yet been systematically evaluated in an randomized control trial (RCT). The proposed study is a one-center, interventional, efficacy study designed to determine antidepressant outcomes of serial ketamine infusions compared to a single ketamine infusion among Veterans with TRD. The investigators have hypothesized that six infusions will be superior to a single infusion of ketamine in both decreasing severity of depressive symptoms and maintaining response. Participants will be male/female Veterans (18 to 75 years old) of any era or military background who suffer from TRD defined as failure to achieve remission from at least 2 antidepressant trials of different pharmacological classes. Potential participants will be recruited from Mental Health clinics and screened for eligibility using a two stage process (phone/chart review, followed by interview). Exclusion criteria includes post-traumatic stress disorder, psychosis-related disorder, bipolar disorder, alcohol/substance use disorder 6 months prior to screening; unstable medical illness; serious/imminent suicidal/homicidal risk; Parkinson's disease, dementia, seizures; traumatic brain injury; contraindicated medications (e.g., MAO inhibitors, barbiturates); received electroconvulsive therapy (ECT) during current episode; pregnancy/nursing. Baseline assessments will be completed 1-2 weeks prior to starting treatment. Participants will be randomly assigned to one of two parallel treatment conditions: 1) six ketamine infusions at 0.5 mg/kg or 2) single ketamine infusion at 0.5 mg/kg preceded by five midazolam infusions at 0.045 mg/kg. Midazolam was chosen as an active placebo given similar pharmacokinetics and dissociative effect profile to ketamine. Each intervention will be provided for a total of 12-day infusion-phase on a Monday-Wednesday-Friday schedule. The, follow-up visits will occur at weekly intervals for the first 4 weeks, at 2-week intervals for the next 8 weeks, and at 4-week intervals for the remaining 12 weeks or until relapse. The primary end point is the Montgomery- sberg Depression Rating Scale (MADRS) score 24 hours following the last infusion where the peak antidepressant effects of ketamine occur. Secondary outcomes for the treatment phase include remission defined by MADRS<10, and response defined as a reduction in the baseline MADRS score 50%. For the follow-up period, durability of antidepressant response will be defined by "time to relapse" to a MADRS score <50% of baseline at that visit. Independent evaluation of depressive symptom severity and potential covariates of antidepressant effect (e.g., pain intensity, level of anxiety) will be ascertained at baseline, at several time points during infusion period, and at follow-up. On the day of infusion, subjects will arrive in the morning after an overnight fast. Hemodynamic measures will be recorded every 10 min for 1 hour beginning 10 min before infusion. Subjects will then receive IV infusion over 40 minutes. Severity of depressive symptoms, pain intensity, level of anxiety will be obtained before and 24 hours after infusion. Acute dissociative effects, manic/hypomanic symptoms, and psychotomimetic effects will be measured 30 minutes before the start of each infusion and at the end of infusion (t0+40 mins) and again at t0+120mins and t0+180mins. The infusion will be discontinued in the event of significant adverse events. Procedures for the subsequent infusions at days 3, 5, 8, 10, and 12 will be identical to those of the first infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veterans aged 18 to 75 years.
* Have a telephone in their home and able to hear telephone conversations.
* Must meet current DSM-IV criteria for major depressive disorder (MDD), single or recurrent, without psychotic features confirmed by depression subset of the Structured Clinical Interview-Clinical Trial for DSM-IV (SCID).
* Have score 32 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30)for severity of major depressive episode (MDE) at screening.
* Current major depressive episode resistant to treatment defined as failure to achieve improvement from at least 2 antidepressant trials of different pharmacological classes. Systematic evaluation of previous antidepressant trials will be assessed by the Antidepressant Treatment History Form (ATHF) .
* If applicable, current antidepressant dosages including augmenting agents and/or frequency and duration of psychotherapy sessions must remain stable for at least 6 weeks prior to beginning of the study.

Exclusion Criteria:

* Inability to speak English.
* Inability or unwillingness to provide written informed consent.
* Moderate/severe cognitive impairment by Mini Mental State Examination (MMSE) scores 27.
* Current or lifetime DSM-V criteria for post-traumatic stress disorder (PTSD), acute stress disorder, psychosis-related disorder, bipolar disorder I or II disorder, substance-induced mood disorder, any mood disorder due to a general medical condition or any Axis I disorder other than MDD as the primary presenting problem.
* History of moderate or severe traumatic brain injury, Parkinson's disease, dementia of any type, multiple sclerosis, seizures or other central nervous system (CNS) related disorders.
* History of comorbid substance disorder within 6 months of assessment plus positive urine toxicology screen test during baseline assessments.
* Clinically unstable medical illness that could compromise the patient's ability to tolerate or likely interfere with the study procedures (e.g., history of or current myocardial ischemia or arrhythmias, congestive heart failure, severe pulmonary, renal, or hepatic disease, uncontrolled hypertension).
* Current or within less than 14 days use of barbiturates or monoamine oxidase inhibitors (MAOi).
* For women: pregnancy (confirmed by lab test), initiation of female hormonal treatments within 3 months of screening, or inability/ unwillingness to use a medically accepted contraceptive method during the study.
* Imminent risk of suicidal/homicidal ideation and/or behavior with intent and/or plan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Shiroma, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shiroma PR, Thuras P, Wels J, Albott CS, Erbes C, Tye S, Lim KO. Neurocognitive performance of repeated versus single intravenous subanesthetic ketamine in treatment resistant depression. J Affect Disord. 2020 Dec 1;277:470-477. doi: 10.1016/j.jad.2020.08.058. Epub 2020 Aug 26. PMID 32871534
- [Result] Shiroma PR, Thuras P, Wels J, Albott CS, Erbes C, Tye S, Lim KO. A randomized, double-blind, active placebo-controlled study of efficacy, safety, and durability of repeated vs single subanesthetic ketamine for treatment-resistant depression. Transl Psychiatry. 2020 Jun 26;10(1):206. doi: 10.1038/s41398-020-00897-0. PMID 32591498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from April 2015 through October 2018
Pre-assignment Details: Four subjects were enrolled but not assigned to treatment. They voluntarily decided to decline participation for logistical issues.
Period: Overall Study
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
Started | 28 | 30
Completed | 25 | 29
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.8) | 51.2 (12.5) | 52.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 22 | 24 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 25 | 46
  Black/African American | 3 | 1 | 4
  Other | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 29 | 54
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
  units on a scale | 34.88 (7.79) | 33.82 (5.11) | 34.32 (6.41)
IDS-C [Mean (Standard Deviation); unit: units on a scale] — The Inventory of Depressive Symptomatology-Clinician Rated (IDS-C) is a 30-item questionnaire designed to assess the severity of depressive symptoms.The seven-day period prior to assessment is the usual time frame for assessing symptom severity. Ranges are 0-11=None, 12-23=Mild, 24-36=Moderate, 37-46=Severe, 47-84=Very Severe.
  units on a scale | 36.8 (3.9) | 39.8 (7.3) | 38.4 (6.1)
BAI [Mean (Standard Deviation); unit: units on a scale] — Beck Anxiety Inventory (BAI) contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. 0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; 26-63: severe anxiety.
  units on a scale | 12.32 (13.62) | 10.57 (6.88) | 11.31 (10.42)
CGI [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 5.32 (0.56) | 5.14 (0.64) | 5.22 (0.60)
NRS [Mean (Standard Deviation); unit: units on a scale] — The NRS for pain is a unidimensional measure of pain intensity in the last 24 hours. An 11-point numeric scale with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable").
  units on a scale | 3.16 (2.49) | 3.37 (2.09) | 3.27 (2.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score After 12 Days of Treatment
Description: Average difference in the Montgomery-Asberg Depression Rating Scale (MADRS) score change between groups. The MADRS has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Time Frame: 13 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
Number analyzed (Participants) | 25 | 29
units on a scale | 21.0 [17.2 to 24.8] | 17.2 [13.2 to 21.2]

2. Secondary Outcome: Antidepressant Response Defined as >50% Decrease in MADRS Baseline Score
Description: Comparing the number of subjects that achieve response between groups as defined above.
Time Frame: 13 days
Measure: Count of Participants; unit: Participants
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
Number analyzed (Participants) | 25 | 29
Participants | 19 | 20

3. Secondary Outcome: Remission Defined as MADRS Score Equal or Less Than 9
Description: Comparing the number of subjects that achieve remission between groups as defined above
Time Frame: 13 days
Measure: Count of Participants; unit: Participants
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
Number analyzed (Participants) | 25 | 29
Participants | 12 | 11

4. Secondary Outcome: Time From Post-infusion Response to Occurrence of Relapse Defined as <50% of Baseline MADRS Score
Description: The length of time from post-infusion response until relapse (defined as >50% of MADRS baseline score) assessed for up to 6 months.
Time Frame: 6 months
Population: The overall number of participants in each intervention corresponds to the total number of subjects that achieve response at the end of six infusions.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
Number analyzed (Participants) | 19 | 20
weeks | 6.00 [0 to 16.81] | 2.00 [0 to 4.92]

ADVERSE EVENTS:
Time Frame: The time frame of data collection was 3 years and 8 months (from April 2015 through December 2018). Each participant was assessed for up to 28 weeks.
Arm/Group | Six Ketamine Infusions | Single Ketamine Infusion Preceded by 5 Midazolam Infusions
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/29
Other Adverse Events (participants affected / at risk) | 17/25 | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Six Ketamine Infusions (N=25) | Single Ketamine Infusion Preceded by 5 Midazolam Infusions (N=29)
Recurrent headaches (Nervous system disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Six Ketamine Infusions (N=25) | Single Ketamine Infusion Preceded by 5 Midazolam Infusions (N=29)
Increased in blood pressure (Cardiac disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 5 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 3
Tremors (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Increased perspiration (Skin and subcutaneous tissue disorders) | 0 | 1
Itching (Skin and subcutaneous tissue disorders) | 1 | 1
Blurred vision (Eye disorders) | 0 | 2
Ringing in ears (Ear and labyrinth disorders) | 0 | 1
Frequent urination (Renal and urinary disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3
Sleeping too much (Nervous system disorders) | 4 | 3
Restlessness (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 5 | 7
Decreased energy (Psychiatric disorders) | 7 | 5
Poor concentration (Nervous system disorders) | 5 | 2
Fatigue (Psychiatric disorders) | 6 | 4
General malaise (General disorders) | 7 | 2
Loss of sexual desire (Reproductive system and breast disorders) | 4 | 3
Trouble achieving orgasm (Reproductive system and breast disorders) | 1 | 2
Trouble with erections (Reproductive system and breast disorders) | 0 | 2
Headaches (Nervous system disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02360280/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02360280/SAP_001.pdf